CLINICAL TRIAL: NCT04355559
Title: Department of Pulmonary & Critical Care Medicine, Chinese PLA General Hospital
Brief Title: The Value of Diaphragmatic Ultrasound in Non-invasive Oxygen Therapy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, wang kaifei, Clinical Professor, Chinese PLA General Hospital
Other Study IDs: 2018TM-03
Record Dates: First submitted 2020-03-24; First posted 2020-04-21 (Actual); Last update posted 2020-04-21 (Actual); Status verified 2020-04

CONDITIONS: Diaphragm Ultrasound; Intensive Care Unit

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- conventional oxygen therapy: Continuous use of current oxygen therapy
- high flow nasal cannula: change the oxygen therapy to high flow nasal cannula
- Noninvasive ventilation: change the oxygen therapy to noninvasive ventilation

SUMMARY:
In this study, a single-center, prospective, observational study was adopted to set the cut-off values of diaphragmatic ultrasound results and arterial blood gas results，with the choice of non-invasive oxygen therapy as the gold standard,so as to evaluate the diagnostic value of diaphragmatic ultrasound in the selection of non-invasive oxygen therapy.

DETAILED DESCRIPTION:
1. the cut-off values of diaphragmatic ultrasound results and arterial blood gas results were established by the selection results of non-invasive oxygen therapy of 120 patients in the intensive care unit and using receiver operating Characteristic curve.

diaphragm excursion，inspiratory time，diaphragm contraction velocity，diaphragm excursion time

ELIGIBILITY:
Inclusion Criteria:

* patients older than 18 years
* without Invasive mechanical ventilation when entering the intensive care unit.

Exclusion Criteria:

* have noninvasive ventilation or high flow nasal cannula contraindications
* history of neuromuscular disease chest wall deformities
* previously assessed diaphragmatic palsy
* shock or severe hemodynamic instability
* known pregnancy, and/or need for immediate endotracheal intubation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients older than 18 years without Invasive mechanical ventilation when entering the intensive care unit.
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2018-08-01 (Actual); Primary Completion 2020-04-30 (Estimated); Study Completion 2020-08-31 (Estimated)

PRIMARY OUTCOMES:
the data diaphragmatic ultrasound | When the intervention which is the first time to change the oxygen therapy
  Record the data at the baseline and intervention

SECONDARY OUTCOMES:
Arterial blood gas analysis results | When the intervention which is the first time to change the oxygen therapy
  Record the data at the baseline and intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Pulmonary and Critical Care Medicine, Chinese PLA General Hospital, Beijing, Beijing Municipality, China